CLINICAL TRIAL: NCT03565575
Title: Improving Risk Perception and Uptake of Pre-exposure Prophylaxis (PrEP) Through Interactive Feedback Based Counselling (and Community Engagement) in Young Women in Manicaland
Brief Title: Manicaland PrEP Uptake Through Interactive Counselling Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Gregson (Other)
Collaborators: Biomedical Research and Training Institute, Zimbabwe (Other); University of Copenhagen (Other); London School of Economics and Political Science (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Simon Gregson, Professor of Demography and Behavioural Science, Imperial College London
Organization: Imperial College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P67251_PrEP; 1R01MH114562-01 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Improving Perceptions of HIV Risk; Improving Uptake of Pre-exposure Prophylaxis for HIV
Keywords: Pre-Exposure Prophylaxis (PrEP) for HIV; Risk perception; HIV

STUDY DESIGN:
Intervention Model Description: matched-cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive tablet-based quiz (Experimental): Individuals participate in an interactive tablet-based risk perception and PrEP counselling information session.
  Interventions: Behavioral: Interactive tablet-based quiz
- Control arm (No Intervention): No intervention will be administered to the control arm

INTERVENTIONS:
Behavioral: Interactive tablet-based quiz — Intervention participants play an interactive tablet based quiz including the following information components:
  1. Risks of HIV infection under different scenarios such as between two hypothetical individuals and with different behaviours.
  2. Interactive counselling on key facts around PrEP, its usability and local availability
  All individuals will have the option to sign up for contact by a nurse from the health clinic to discuss PrEP further and make an appointment for a visit. Participants will also be given a PrEP referral letter which they can present directly at one of the participating study clinics to begin PrEP. In two sites a community-led intervention will also be implemented to address social obstacles and to increase support from peers, families and social structures.
  Arms: Interactive tablet-based quiz

SUMMARY:
Primary Objective:

The purpose of this trial is to evaluate the impact of an interactive tablet based counselling session correcting risk perception and addressing ambiguity around availability, usability and effectiveness of PrEP on PrEP uptake within 6 months in adolescent girls and young women (AGYW) aged 18-24 years.

Hypothesis:

Correcting misperceptions of risks of HIV infection and off-setting ambiguity effects about the availability, usability and efficacy of PrEP, through localized, interactive, tablet-based counselling, will increase uptake of PrEP in HIV-negative AGYW.

Study outcomes:

The primary outcomes for the study will be risk perception measured in a follow-up survey at 6 months and proportion of women taking up PrEP within 6 months measured with biomarkers of plasma antiretroviral (ARV) drug presence.

DETAILED DESCRIPTION:
With 6 clusters per arm, mean cluster size of 48 individuals, with co-efficient of variation in outcomes between 0.15 to 0.55, the trial will have 80% power to detect difference of 5 - 9 percentage points when baseline PrEP uptake is assumed to be 1%.

Primary analysis:

A two-stage intention-to-treat (ITT) analysis of cluster level summaries will be used. The parameter of interest is the adjusted risk difference in primary and secondary outcomes.

In the first stage, Logistic regression will be used to adjust for confounding variables at the individual level. The model will be fitted using data from both trial arms. The regression model will include terms for the covariates of interest and pair but not trial arm. Adjustment variables will include age group (<20, 20-24), highest level of education completed, marital status and baseline measures of outcomes. In the second stage, a formal statistical comparison for differences in observed versus expected uptake by arm will be conducted using a two-sided paired significance test with α=0.05.

Secondary analysis:

In secondary analysis, the complier average causal effect (CACE) will be estimated using an instrumental variables approach. The parameter of interest is the adjusted risk difference in primary and secondary outcomes.

Heterogeneity by age and baseline levels of risk and time preferences will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-24 years

Exclusion Criteria:

* Participants testing HIV-positive at baseline
* Self-reporting taking PrEP at baseline

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 1055 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Uptake of Pre-exposure prophylaxis for HIV | 6 months
  The proportion of women taking up PrEP within 6 months measured with biomarkers of plasma ARV presence.

SECONDARY OUTCOMES:
Changes in perception of risk of HIV from age-disparate partnerships | 6 months
  Risk perception with be measured in a follow-up survey at 6 months with the following specific definitions
  * Proportion of women correctly reporting a 25-29 year old man is more likely infected with HIV in Manicaland than a 15-19 year old man
  * Proportion of women correctly reporting a 25-29 year old man is more likely infected with HIV in Manicaland than a 15-19 year old woman

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gregson, PhD, Principal Investigator — Imperial College London
Locations (8):
- Zimbabwe (8):
  - Manicaland Centre for Public Health Research, Bonda, Manicaland Province
  - Manicaland Centre for Public Health Research, Eastern Highlands, Manicaland Province
  - Manicaland Centre for Public Health Research, Hobhouse, Manicaland Province
  - Manicaland Centre for Public Health Research, Honde, Manicaland Province
  - Manicaland Centre for Public Health Research, Nyazura, Manicaland Province
  - Manicaland Centre for Public Health Research, Sakubva, Manicaland Province
  - Manicaland Centre for Public Health Research, Selbourne, Manicaland Province
  - Manicaland Centre for Public Health Research, Nyanga

REFERENCES:
- [Derived] Thomas R, Skovdal M, Galizzi MM, Schaefer R, Moorhouse L, Nyamukapa C, Maswera R, Mandizvidza P, Hallett TB, Gregson S. Improving risk perception and uptake of pre-exposure prophylaxis (PrEP) through interactive feedback-based counselling with and without community engagement in young women in Manicaland, East Zimbabwe: study protocol for a pilot randomized trial. Trials. 2019 Dec 2;20(1):668. doi: 10.1186/s13063-019-3791-8. PMID 31791405